CLINICAL TRIAL: NCT02704286
Title: Raising Awareness of Knee Osteoarthritis (OA) and Willingness to Undertake Behavioral Changes to Reduce Risk of Knee OA: Online Recruitment
Brief Title: Risk and Risk Perception of Knee Osteoarthritis in the US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elena Losina, Professor of Orthopedic Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015P000249
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic Osteoarthritis Risk Information (Sham Comparator): Participants in this arm received generic osteoarthritis information that was not personalized.
  Interventions: Behavioral: Generic osteoarthritis information
- Personalized Osteoarthritis Risk (Experimental): Participants in this arm obtained their personalized osteoarthritis risk from the internet-based Osteoarthritis Risk Calculator.
  Interventions: Behavioral: Internet-Based Osteoarthritis Risk Calculator

INTERVENTIONS:
Behavioral: Internet-Based Osteoarthritis Risk Calculator — The investigators have developed a personalized risk calculator for knee osteoarthritis. This risk calculator uses the Osteoarthritis Policy Model to estimate an individual's risk of developing knee osteoarthritis within their lifetime based on demographic information and risk factors. It shows this information to the user with interactive graphs and compares their risk to the risk of an average American of the same age.
  Arms: Personalized Osteoarthritis Risk
Behavioral: Generic osteoarthritis information — Subjects viewed generic (i.e. not personalized) information about osteoarthritis risk factors
  Arms: Generic Osteoarthritis Risk Information

SUMMARY:
The investigators have created an interactive knee osteoarthritis (OA) risk calculator that estimates a user's risk of developing symptomatic knee OA as well as the user's risk for undergoing a total knee replacement (TKR) within their lifetime. To test the impact of the calculator, the investigators recruited OA-free subjects from Amazon's Mechanical Turk. Participants were randomized to either access general information about OA or use the risk calculator in addition to accessing general OA information. The investigators hypothesized that participants randomized to the risk calculator arm would have more accurate perception of their knee OA risk and would have increased willingness to change risky behavior compared to the general OA information group.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 25 and 45
* Participants must live in the United States
* Participants must not be diagnosed with osteoarthritis

Exclusion Criteria:

* All participants who did not meet the inclusion criteria

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in estimated lifetime knee OA risk | 1 day
  The difference between average lifetime knee osteoarthritis risk estimated by participants at baseline and average lifetime knee osteoarthritis risk estimated by participants after the intervention.
Change in estimated 10-year knee OA risk | 1 day
  The difference between average 10-year knee osteoarthritis risk estimated by participants at baseline and average 10-year knee osteoarthritis risk estimated by participants after the intervention.

SECONDARY OUTCOMES:
Reaching an Action Stage on Diet Contemplation Ladder | 1 day
  The percentage of subjects who originally ranked themselves below an action stage (8 or higher) on a contemplation ladder for changing diet related behaviors and who moved to an action stage after the intervention.
Reaching an Action Stage on Exercise Contemplation Ladder | 1 day
  The percentage of subjects who originally ranked themselves below an action stage (8 or higher) on a contemplation ladder for changing exercise related behaviors and who moved to an action stage after the intervention.
Reaching an Action Stage on Weight Control Contemplation Ladder | 1 day
  The percentage of subjects who originally ranked themselves below an action stage (8 or higher) on a contemplation ladder for changing weight control behaviors and who moved to an action stage after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Losina, PHD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Losina E, Klara K, Michl GL, Collins JE, Katz JN. Development and feasibility of a personalized, interactive risk calculator for knee osteoarthritis. BMC Musculoskelet Disord. 2015 Oct 22;16:312. doi: 10.1186/s12891-015-0771-3. PMID 26494421
- [Background] Michl GL, Katz JN, Losina E. Risk and risk perception of knee osteoarthritis in the US: a population-based study. Osteoarthritis Cartilage. 2016 Apr;24(4):593-6. doi: 10.1016/j.joca.2015.11.001. Epub 2015 Nov 7. PMID 26555504
- [Derived] Losina E, Michl GL, Smith KC, Katz JN. Randomized Controlled Trial of an Educational Intervention Using an Online Risk Calculator for Knee Osteoarthritis: Effect on Risk Perception. Arthritis Care Res (Hoboken). 2017 Aug;69(8):1164-1170. doi: 10.1002/acr.23136. Epub 2017 Jul 10. PMID 27788299